CLINICAL TRIAL: NCT07177898
Title: ALLOPURINOL AND LISINOPRIL FOR DIABETIC KIDNEY PROTECTION: A COMPARATIVE STUDY IN NORMOURICEMIC TYPE 2 DIABETICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Narowal Medical College (Other Government)
Collaborators: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Sami Ullah Mumtaz, Associate Professor, Narowal Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 163/RC/KEMU
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Kidney Disease (DKD)
Keywords: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A received allopurinol with lisinopril
  Interventions: Drug: Allopurinol
- Group B (No Intervention): Group B received Lisinopril alone

INTERVENTIONS:
Drug: Allopurinol — Group A received allopurinol with lisinopril, and Group B received lisinopril alone
  Arms: Group A

SUMMARY:
This randomized controlled trial was conducted at the Department of Medicine and Diabetes of Mayo Hospital/King Edward Medical University, Lahore, over one year. A total of 80 patients with type 2 diabetes and normal serum uric acid were randomly assigned to two groups: Group A received allopurinol with lisinopril, and Group B received lisinopril alone. Patients were monitored every three months for serum creatinine, spot urine albumin, and serum uric acid levels. The primary endpoint was a >300 mg/L increase in urine albumin from baseline. Blood pressure was managed with agents other than ACE inhibitors if required.

DETAILED DESCRIPTION:
This study is a randomized controlled trial conducted at the Department of Medicine and the Diabetic Clinic of Mayo Hospital/King Edward Medical University, Lahore. The duration of the study was one year, starting from the acceptance of the research synopsis. The estimated sample size was 80 patients (40 in each group), calculated using a 5% level of significance, a 90% power of the test and expected percentages of 84% for the allopurinol group and 54% for the placebo group. Probability simple random sampling was used for patient selection. Inclusion criteria for the study included patients with type 2 diabetes mellitus on oral hypoglycemic agents, serum creatinine levels less than 1.1 mg/dL, and serum uric acid levels between 5.5-6.5 mg/dL for males and 5-6 mg/dL for females. Additionally, patients must be over the age of 35 and from both genders. Exclusion criteria included patients with tumor lysis syndrome, chronic kidney disease from other causes (e.g., hypertension, glomerulonephritis, polycystic kidney disease, or hydronephrosis), those on medications that could cause hyperuricemia (such as thiazide diuretics) or those on drugs that may induce proteinuria (e.g., NSAIDs, cyclosporine, penicillamine, or gold). Patients with uric acid levels exceeding 7 mg/dL were also excluded. A total of 80 patients who met the inclusion criteria were selected from the outpatient department of medicine and the diabetic clinic. Informed consent was obtained from all participants prior to the intervention. Demographic data, including the duration of diabetes diagnosis, were recorded. Patients were randomly assigned to one of two groups via a lottery method: Group A received allopurinol in combination with lisinopril therapy, and Group B received lisinopril therapy alone. Over the course of one year, all patients were monitored every three months for serum creatinine, spot urine albumin levels, and serum uric acid levels. An increase in urine albumin levels by more than 300 mg/L from baseline was considered the endpoint. If a patient developed uncontrolled hypertension during the study, the dose of ACE inhibitors (lisinopril) was not increased beyond 5 mg; instead, additional antihypertensive agents were used to manage blood pressure. Data analysis was performed using SPSS-20, with quantitative variables such as age presented as mean ± SD and qualitative variables such as sex presented as frequency and percentage. To compare the progression of nephropathy between the allopurinol and placebo groups, an independent sample t-test was applied, with p-values ≤ 0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes mellitus on oral hypoglycemic agents, serum creatinine levels less than 1.1 mg/dL, and serum uric acid levels between 5.5-6.5 mg/dL for males and 5-6 mg/dL for females

Exclusion Criteria:

* patients with tumor lysis syndrome, chronic kidney disease from other causes (e.g., hypertension, glomerulonephritis, polycystic kidney disease, or hydronephrosis), those on medications that could cause hyperuricemia (such as thiazide diuretics) or those on drugs that may induce proteinuria (e.g., NSAIDs, cyclosporine, penicillamine, or gold). Patients with uric acid levels exceeding 7 mg/dL were also excluded

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-14 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Urinary Albumin | 3 months
  The primary endpoint was a >300 mg/L increase in urine albumin from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
I do not have the permission of my institute to share the date under the sanctity of data.

REFERENCES:
- [Background] Robinson RL, et al. Allopurinol reduces proteinuria in diabetic nephropathy: A randomized controlled trial. Diabetologia. 2020;63(6):1217-1224.